CLINICAL TRIAL: NCT00111072
Title: Dexamethasone 0.01% Solution for the Treatment of Oral Lichen Planus
Brief Title: Dexamethasone to Treat Oral Lichen Planus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050155; 05-D-0155
Record Dates: First submitted 2005-05-16; First posted 2005-05-16 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2006-03

CONDITIONS: Oral Lichen Planus
Keywords: Mucosal Disease; Topical Steroids; Salivary Diagnostics; Oral Pain; Quality of Life Indicators; Oral Lichen Planus
MeSH Terms: conditions — Lichen Planus, Oral | interventions — Dexamethasone; Solutions

INTERVENTIONS:
Drug: dexamethasone 0.01% solution

SUMMARY:
This study will evaluate the effectiveness of dexamethasone 0.01% solution in treating pain associated with oral lichen planus, a chronic disease that causes painful ulcers inside the mouth. The cause of lichen planus not known, but it may be related to an allergic or immune reaction. This study will examine what causes the disease, the pain associated with it, its impact on patients' lives and the use of dexamethasone to treat it.

Patients 12 or older with severe oral lichen planus may be eligible for this study. Candidates are screened with blood tests and a biopsy to confirm the diagnosis and provide tissues for research purposes. For the biopsy, two small circles of tissue, each about 4 mm (1/5 inch) across, are surgically removed.

Participants are randomly assigned to rinse their mouth with either a dexamethasone solution or placebo (a rinse with no active ingredient) four times a day for 4 weeks. During this period they may not use any oral or topical pain or anti-inflammatory medications except diphenhydramine 12.5 mg/5 ml (a topical numbing medicine) and Tylenol, both which are provided by the study.

Patients come to the NIH Clinical Center for three 1-hour visits (once every two weeks) and once more 4 weeks after the study medications are stopped. At the first three visits patients submit a pain diary in which they have recorded information on pain levels, and they are checked for any medication side effects. On the third visit (the last day they take the study drug) they are also tested for adrenal suppression that may have resulted from taking the steroid rinse. For this test they are given an injection of a drug called synacthen and after 1 hour, a blood sample is drawn. Patients return for a final visit 1 month later to determine if their disease returns or improves after the medication is stopped.

DETAILED DESCRIPTION:
This is a study of pain, oral function and salivary biomarkers in oral lichen planus.

The primary objective of the study is to determine the efficacy of dexamethasone rinse in reducing pain in patients with oral lichen planus. Secondary objectives are to evaluate a novel scoring system of severity of lichen planus, assess the changes in salivary biomarkers associated with the treatment, assess the impact of oral lichen planus on the quality of life using the SF-36 instrument and the Oral Health Impact Profile (OHIP-14).

This is a double-blind parallel group design with 20 patients in each arm. Our primary outcome measure will be change in the visual analog scale that assesses pain. We will consider a decrease of 30 mm as clinically significant. Secondary outcomes will include reduction of oral symptoms as measured by the OHIP-14, amount of topical analgesic used, improvement in quality of life scores, and the severity of lesions as assessed with two scales.

A new oral lichen planus scoring system will be evaluated for validity, reliability and sensitivity to change. This system will quantify the severity and amount of oral lichen planus lesions on a scale of 0 to 66. Validation of this scale is needed for future studies of oral lichen planus. The validity and sensitivity to change will be assessed by correlation of the scores with patient based outcomes as well as global scale. Inter- and intra-rater reliability will also be tested.

The principal study interventions will be dexamethasone 0.01% oral rinse or identical in appearance and taste placebo rinse. Additional allowed interventions will be standard oral topical analgesic rinse and acetaminophen on an as needed basis. Diagnostic and research evaluations will include complete history and oral and general physical examination, laboratory investigations, saliva collection, and oral mucosal biopsy. The interventional period of the trial will be 4 weeks.

ELIGIBILITY:
INCLUSION CRITERIA:

Biopsy confirmed symptomatic oral lichen planus. World Health Organization histological criteria (12) in combination with a compatible clinical appearance will be used for diagnosis.

No current treatment with immunomodulatory agents. A one-month washout period will be required prior to enrollment if patients are taking immunomodulatory agents. Prior treatment with topical steroids will be allowed provided the presence of symptomatic lesions.

Age greater than 12 years old. Lichen planus is very rare in patients younger than 40 years old. Patients must rinse and spit the medication rather than swallow it. Oral rinses such as topical fluorides are not recommended for young children.

Patients of both sexes and all racial and ethnic groups will be eligible.

Symptomatic lichen planus with a score of at least 35 mm on a visual analog scale for pain.

Oral lichen planus score of at least 3 on the lichen planus severity scale.

EXCLUSION CRITERIA:

Unable to undergo oral biopsy for diagnosis.

Asymptomatic lichen planus with no ulcerated or erythematous oral lesions.

Treatment with immunomodulatory agents within 1 month of the randomization.

Hepatitis C infection.

Documented hypersensitivity to dexamethasone.

Pregnancy or lactation.

Poorly controlled diabetes.

Inability or unwillingness to give written informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70
Dates: Start 2005-05; Study Completion 2006-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Dental And Craniofacial Research (NIDCR), Bethesda, Maryland, United States

REFERENCES:
- [Background] Axell T, Rundquist L. Oral lichen planus--a demographic study. Community Dent Oral Epidemiol. 1987 Feb;15(1):52-6. doi: 10.1111/j.1600-0528.1987.tb00480.x. PMID 3467894
- [Background] Eisen D. The clinical manifestations and treatment of oral lichen planus. Dermatol Clin. 2003 Jan;21(1):79-89. doi: 10.1016/s0733-8635(02)00067-0. PMID 12622270
- [Background] Scully C, Beyli M, Ferreiro MC, Ficarra G, Gill Y, Griffiths M, Holmstrup P, Mutlu S, Porter S, Wray D. Update on oral lichen planus: etiopathogenesis and management. Crit Rev Oral Biol Med. 1998;9(1):86-122. doi: 10.1177/10454411980090010501. PMID 9488249